CLINICAL TRIAL: NCT04165044
Title: Leucocytes - and Platelet Rich Fibrin Versus Connective Tissue Graft Associated to Coronally Advanced Flap in the Treatment of Miller Class I and II Localized Gingival Recession: A Randomized Controlled Clinical Trial
Brief Title: L-PRF Versus Connective Tissue Graft Associated to Coronally Advanced Flap in Gingival Recession Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Catherine Andrade, Principal investigator, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L-PRF in gingival recession
Record Dates: First submitted 2019-11-07; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Gingival Recession, Localized
Keywords: Leukocyte and Platelet Rich Fibrin; Connective tissue graft; Gingival recession
MeSH Terms: conditions — Gingival Recession | interventions — Leukocyte Count

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial of parallel group (1:1)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The clinician who performed the measurements as well as the statistic were blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF+CAF (Active Comparator): Leukocyte and Platelet Rich Fibrin plus Coronally Advanced Flap
  Interventions: Procedure: Leukocyte and Platelet Rich Fibrin plus Coronally Advanced Flap
- CTG+CAF (Active Comparator): Connective Tissue graft plus Coronally Advanced Flap
  Interventions: Procedure: Connective tissue graft plus Coronally Advanced Flap

INTERVENTIONS:
Procedure: Leukocyte and Platelet Rich Fibrin plus Coronally Advanced Flap — The Coronally advanced flap was made following the protocol described by Zucchelli et al. in 2007. (39). When the margin of the flap was able to passively extend until more coronal of the CEJ the coronal mobilization of the flap was considered satisfactory. A double L-PRF membrane was positioned at the level of CEJ, getting the stabilization with 5-0 resorbable suture. After that, the flap was coronally advanced and stabilized with interrupted sutures (5-0 resorbable) anchored to incisal contact points (mesial and distal) created with a flowable, light-curing resin material in the treated tooth. Finally, gentle pressure over the area with a moistened gauze with saline solution was performed.
  Other Names: L-PRF + CAF
  Arms: L-PRF+CAF
Procedure: Connective tissue graft plus Coronally Advanced Flap — The Coronally advanced flap was made following the protocol described by Zucchelli et al. in 2007. (39). When the margin of the flap was able to passively extend until more coronal of the CEJ the coronal mobilization of the flap was considered satisfactory. Then connective tissue graft obtained from the palate was positioned at the level of CEJ, getting the stabilization with 5-0 resorbable suture. After that, the flap was coronally advanced and stabilized with interrupted sutures (5-0 resorbable) anchored to incisal contact points (mesial and distal) created with a flowable, light-curing resin material in the treated tooth. Finally, gentle pressure over the area with a moistened gauze with saline solution was performed.
  Other Names: CTG + CAF
  Arms: CTG+CAF

SUMMARY:
Background: Nowadays, the use of connective tissue graft associated to the coronally advanced flap is considered the "gold standard" for localized gingival recession treatment. However, this technique requires a donor site, which can be associated with greater morbidity. The use of platelet concentrates, particularly the Leukocytes- and Platelets Rich Fibrin (L-PRF), it has emerged as an alternative for gingival recession treatment, due to its properties which enhance the regenerative process. Therefore, the purpose of this study was to evaluate and to compare the effect obtained with L-PRF versus connective tissue graft (CTG) associated to the Coronally Advanced Flap (CAF) in the treatment of Miller class I or II localized gingival recessions.

Methods: A randomized controlled clinical trial of parallel groups (1:1) with 17 recessions in each group was performed. Control group (CAF + CTG) and test group (CAF + L-PRF). In each group the following variable were measured: postoperative pain and incidence of post-surgical complications at 24-48-72 hours, gingival recession depth (RD), gingival recession width (RW), gingival thickness (GT), probing depth (PD), clinical insertion level (NIC), keratinized tissue height (KTH) before treatment and after 1, 3 and 6 months of root covering surgery and the root coverage esthetic score (RES) at 6 months after treatment.

DETAILED DESCRIPTION:
Study design and participants A randomized controlled clinical trial of parallel groups (1:1) with 17 recessions in each group was performed. Control group (CAF + CTG) and test group (CAF + L-PRF). This study was approved by the ethical committee of Universidad de Los Andes, Santiago Chile (CEC201627) and in full accordance with the ethical principles of the Declaration of Helsinki, as revisited in 2000. The patients were instructed about the benefits and risks of the study and each participant signed an informed consent form.

Thirteen patients (9 females and 4 males; aged 26 to 53 years; mean year: 41,74; SD: 9,11 years) with a total of 34 gingival recession (27 in females and 7 in males) participated in the present study. (Figure 1)

The sample size was based on the detection of 1 mm difference in gingival recession reduction between the treatment groups (standard deviation 0.93), with a two-sided 5% significance level, a power of 85%.(36) The sample size calculation was obtained using the software STATA v14.0.

Initial therapy and clinical measurements The patient enrolled received a prophylaxis session (scaling and professional tooth cleaning), all patients had less of 20% of plaque or 80% oral hygiene according to the O´Leary oral hygiene index.(37) All clinical parameters measurements were performed by a single trained and calibrated examiner (C.A.) and masked for the treatment assigned. An Individual acrylic stents were prepared for all patients to take measurements of the constant points.

The following parameters were evaluated at baseline and 1, 3, and 6 months after treatment: 1) gingival recession depth (RD), distance between CEJ and gingival margin (GM); 2) gingival recession wide (RW), measured at CEJ level; 3) probing depth (PD), measured from margin of the gingiva to the gingival sulcus base; 4) clinical attachment level (CAL), measured from the CEJ to the gingival sulcus base; 5) keratinized tissue height (KTH), measured from the mucogingival junction to the gingival margin; 6) gingival thickness (GT) at 3 mm from the gingival margin, measured un local anesthesia with an endodontic spacer Nº 25 with its stopper silicone disc and an endodontic rule; 7) root coverage (RC) was calculated in millimeters and percentages according to the following formula: [(pre-operative RD - post-operative RD)/pre-operative RD] × 100.

PD, CAL, and KTH measurements were performed at the mid-buccal aspect of the teeth, by a manual probe and were rounded up to the nearest millimeter.(7)

Patient Evaluation of Postoperative Morbidity and Esthetics Pain score using a 100-mm visual analogue scale (VAS) (0 indicating no pain, 50 indicating average, and 100 indicating an unbearable pain) and the incidence of complications post-surgery (such as hematoma, swelling, bleeding, infection, wound dehiscence, etc.) responding dichotomous questions, were registered at 24, 48 and 72 hours after the surgery.

The root coverage esthetic score (RES) was evaluated at 6 months according to the protocol of Cairo et al.(38).

Surgical treatment Prior to starting the surgery, the surgeon opened the envelope labeled with the assigned treatment. All surgeries were performed by a single expert periodontist (A.S.). Under local anesthesia, the root area corresponding to buccal attachment loss (gingival recession + buccal PD) was instrumented with Gracey curettes until obtain a polished surface. Then, the surface was washed with a saline solution for 30 seconds. Additionally, a chemical treatment of the root surface for 3 minutes was done using Tetracycline HCl (250 mg/ml), mixing 250 mg in 1 ml of sterile water. After that, the root surface was rinsed for 60 seconds with saline solution.

The CAF was made following the protocol described by Zucchelli et al. in 2007. (39). Two horizontal beveled incision were done at mesial and distal of the gingival recession (each one 3 mm in length) at a distance from the tip of the anatomical papillae equal to the depth of the recession plus 1 mm. Both incisions were connected with an intrasulcular incision. From the horizontal incisions, two beveled obliques, slightly divergent, incisions were extended until the alveolar mucosa. Then, the trapezoidal-shaped flap, split-full-split from coronal to apical was elevated and the papillae (mesial and distal) were deepithelialized. When the margin of the flap was able to passively extend until more coronal of the CEJ the coronal mobilization of the flap was considered satisfactory.

According to the treatment assignment (control or test group), a connective tissue graft or a double L-PRF membrane was positioned at the level of CEJ, getting the stabilization with 5-0 resorbable suture. After that, the flap was coronally advanced and stabilized with interrupted sutures (5-0 resorbable) anchored to incisal contact points (mesial and distal) created with a flowable, light-curing resin material in the treated tooth. Finally, a gentle pression over the area with a moistened gauze with saline solution was performed.

L-PRF preparation 2 vacutainer tubes of 10 ml without anticoagulant of blood were obtained and centrifuged at 408 g for 12 minutes using a table centrifuge (IntraSpinTM, Intralock, Florida, USA) according to the protocol described by Temmerman et al. in 2016.(40) The L-PRF clots obtained were removed from the tube, separated of the red cells and located inside of Xpression box (IntraSpinTM, Intralock, Florida, USA) to convert them into membranes.

The two L-PRF membranes obtained were attached using a resorbable suture until obtain only one thicker and stable membrane. (Figure 2)

Postsurgical indications and control pain Ketoprofen 100 mg was administrated immediately before the surgery. Then, they took the same prescription every 12 hours for the next 2 days. In some specific cases, the prescription was extended to control pain and the extra doses was registered.

The patients received written and oral instructions about not touch the involved area, only liquid diet and do not make any hard effort or sports activity during two weeks until the sutures were removed. Related to oral hygiene after surgery, the patients were also instructed to not brush their treated teeth, just rinse with Chlorhexidine solution (0.12%) three times a day for 1 min. After suture removal, the chlorhexidine rinsing was maintained for additional 2 weeks. After that, the patients were again instructed with a -traumatic tooth brushing technique.

Randomization, Allocation Concealment, and Calibration Computer-Generated randomization was used to assign the patients with an allocation ratio of 1:1 into two study groups: CAF + L-PRF (17 gingival recession; control) and CAF + CTG (17 gingival recession; test). To conceal the treatment assignment, opaque envelopes containing the name of the intervention were used. During the intra-examiner calibration period, a 90% level of calibration (K coefficient = 0.90) was detected after triplicate measurement of gingival recession depth (GRD), distance from the CEJ to the margin of the gingiva, in 50 recession defects.

Statistical analysis Descriptive analysis was expressed as mean and standard deviation (SD) or median and interquartile range (IQR) according to distribution of data (normality) determinate by Shapiro-Wilk test. Student's t-test was used to evaluate differences between baseline measures and different evaluations times of variables expresses as mean, in the variables expresses as median was used the Wilcoxon test was applied. Categorical measurement was analyzed by Chi-square test. A p-value < 0.05 considered as significant in all tests. The analysis was performed with Stata software v.12, Stata Corp, College Station, TX.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients
* Older than18 years
* At least one localized Miller class I or II gingival recession higher than 3mm at buccal aspect of anterior/premolar area
* An identifiable cement-enamel junction (CEJ)
* Without bleeding on probing (BOP)
* Pulp vitality

Exclusion Criteria:

* Smokers
* Pregnancy
* Active periodontal disease
* Previous periodontal surgical procedures in the recession area
* Coagulation disorders
* Anticoagulant treatment
* Patients who cannot comply the study and/or maintenance visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Recession depth (RD) | At 1 month, 3 months and 6 months
  pre-operative RD - post-operative RD in millimeters

SECONDARY OUTCOMES:
Change in Recession wide (RW) | At 1 month, 3 months and 6 months
  pre-operative RW - post-operative RW in millimeters
Change in Percentage of root coverage | At 1 month, 3 months and 6 months
  [(pre-operative RD - post-operative RD)/pre-operative RD] × 100 = (%)
Change in Gingival thickness (GT) | At 1 month, 3 months and 6 months
  pre-operative GT - post-operative GT in millimeters
Change in Probing depth (PD) | At 1 month, 3 months and 6 months
  pre-operative PD - post-operative PD in millimeters
Change in Clinical attachment level (CAL) | At 1 month, 3 months and 6 months
  pre-operative CAL - post-operative CAL in millimeters
Change in Keratinized tissue height (KTH) | At 1 month, 3 months and 6 months
  pre-operative KTH - post-operative KTH in millimeters
Post- operative pain | At 24, 48 and 72 hours after surgery.
  Mean of Visual Analogue Scale score . Outcomes from: no pain (0 mm) until severe pain (maximum 100 mm).
Root Coverage Esthetic Score (RES) | At 6 months
  Mean of Root Coverage Esthetic Score. Outcomes: from 0 (worse outcome) until 10 (better outcome)
Post-surgery complications incidence | At 24, 48, 72 hours.
  Frequency and percentage of post-surgery complications

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Andrade, Principal Investigator — Universidad de Los Andes
Locations (1):
- Universidad de Los Andes, Santiago, Chile